CLINICAL TRIAL: NCT03745989
Title: Phase 1b Open-label Study of MK-8353 in Combination With Selumetinib (MK-5618) in Participants With Advanced/Metastatic Solid Tumors
Brief Title: Study of MK-8353 + Selumetinib in Advanced/Metastatic Solid Tumors (MK-8353-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8353-014; MK-8353-014 (Other: Merck)
Record Dates: First submitted 2018-11-16; First posted 2018-11-19 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Solid Tumors
Keywords: advanced/metastatic; solid tumors; Selumetinib
MeSH Terms: conditions — Neoplasm Metastasis | interventions — MK-8353; AZD 6244

STUDY DESIGN:
Intervention Model Description: Groups of participants are assigned to receive interventions based on prior milestones being reached in the study, such as in some dose escalation and adaptive design studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-8353 and Selumetinib Dose Escalation (Experimental): Participants will receive a combination MK-8353 and selumetinib for 4 days on and 3 days off until disease progression or discontinuation. MK-8353 will be escalated sequentially from 50 mg to 250 mg based on pharmacokinetic and safety data. Selumetinib will be escalated sequentially from 25 mg to 75 mg based on pharmacokinetic and safety data. Doses may be adjusted downward sequentially based on tolerability
  Interventions: Drug: MK-8353; Drug: Selumetinib

INTERVENTIONS:
Drug: MK-8353 — Participants will receive MK-8353 orally twice daily (BID), escalated sequentially from 50 mg to 250 mg.
Drug: Selumetinib — Participants will receive selumetinib orally BID, escalated sequentially from 25 mg to 75 mg.
  Other Names: MK-5618

SUMMARY:
This is a multicenter, worldwide, open-label study of MK-8353 in combination with selumetinib in participants with histologically or cytologically confirmed diagnosis of advanced solid tumor. This study will evaluate the safety, tolerability, and exploratory efficacy of MK-8353 in combination with selumetinib.

DETAILED DESCRIPTION:
As specified by Phase 1 protocol-flexible language, modifications to the dose or dosing regimen can be made to achieve the scientific goals of the trial objectives and/or ensure appropriate safety of the trial participants. The proposed doses may be adjusted based on evaluation of safety, tolerability, and pharmacokinetic data.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically- or cytologically-documented, locally-advanced or metastatic solid tumor by pathology report and have received, or been intolerant to, all treatment known to confer clinical benefit.
* Provide an archival or newly obtained tumor tissue sample and blood samples for assessment of proto-oncogene rat sarcoma virus (RAS)/rapidly accelerated fibrosarcoma (RAF) mutation and for biomarker analysis.
* Have at least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) on imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) as assessed by the investigator/local radiology review.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale. (Obtain within 7 days prior to first dose of study treatment.)
* Have the ability to swallow and retain oral medication.
* Demonstrate adequate organ function.
* Male participants must agree to use an acceptable contraception during the treatment period and for at least 120 days after the last dose of study intervention and refrain from donating sperm during this period.
* Female participants must not be pregnant, not breastfeeding, and either not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the study's contraceptive guidance during the treatment period and for at least 120 days, after the last dose of study intervention.

Exclusion Criteria:

* Have had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) prior to the first dose of study treatment, or has not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from any AEs that were due to cancer therapeutics administered more than 4 weeks earlier (this includes participants with previous immunomodulatory therapy with residual immune-related AEs).
* Have clinically active central nervous system metastases and/or carcinomatous meningitis.
* Have an active infection requiring therapy.
* Have known human immunodeficiency virus (HIV) and/or Hepatitis B or C infections, or known to be positive for Hepatitis B antigen (HBsAg)/ Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) or Hepatitis C Antibody or ribonucleic acid (RNA).
* Have clinically significant cardiovascular disease as defined by study criteria.
* Have a history of thromboembolic or cerebrovascular events within 6 months prior to treatment start, including transient ischemic attacks (TIAs), cerebrovascular accidents (CVAs), deep vein thrombosis, or pulmonary embolism.
* Have neuromuscular disorders associated with an elevated creatine kinase (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Have one or more study-defined ophthalmological findings/conditions.
* Have a known history of Gilbert's Syndrome.
* Have a history or current evidence of a gastrointestinal (GI) condition (e.g., inflammatory bowel disease, Crohn's disease, ulcerative colitis) or impaired liver function or diseases that in the opinion of the investigator may significantly alter the absorption or metabolism of oral medications.
* Have a known psychiatric or substance abuse disorder, or any other cognitive disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the Screening Visit through 120 days after the last dose of study treatment.
* Received prior therapy with a mitogen activated protein kinase (MEK) inhibitor (e.g., cobimetinib, trametinib), or an extracellular signal-regulated kinase (ERK) inhibitor (e.g., MK-8353, GCD-0994, ulixertinib), or a proto-oncogene BRAF inhibitor (e.g., dabrafenib, vemurafenib).
* Is currently participating and receiving study treatment in a study of an investigational agent or has participated and received study treatment in a study of an investigational agent or has used an investigational device within 28 days of administration of selumetinib.
* Have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to agents and/or excipients used in the study.
* A WOCBP who has a positive urine pregnancy test within 24 hours before the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- United States (2):
  - Florida Cancer Specialists ( Site 7000), Sarasota, Florida
  - Next Oncology ( Site 0001), San Antonio, Texas
- Canada (2):
  - BC Cancer-Vancouver Center ( Site 0011), Vancouver, British Columbia
  - Princess Margaret Cancer Centre ( Site 0012), Toronto, Ontario
- Istituto Oncologica della Svizzera Italiana (IOSI) ( Site 0020), Bellinzona, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Stathis A, Tolcher AW, Wang JS, Renouf DJ, Chen LC, Suttner LH, Freshwater T, Webber AL, Nayak T, Siu LL. Results of an open-label phase 1b study of the ERK inhibitor MK-8353 plus the MEK inhibitor selumetinib in patients with advanced or metastatic solid tumors. Invest New Drugs. 2023 Jun;41(3):380-390. doi: 10.1007/s10637-022-01326-3. Epub 2023 Apr 11. PMID 37040046
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-8353 50 mg + Selumetinib 25 mg: Participants received 50 mg twice daily (BID) of MK-8353 and 25 mg selumetinib orally with 4 days on and 3 days off until disease progression or discontinuation.
- MK-8353 100 mg + Selumetinib 50 mg: Participants received 100 mg BID of MK-8353 and 50 mg selumetinib orally with 4 days on and 3 days off until disease progression or discontinuation.
- MK-8353 150 mg + Selumetinib 75 mg: Participants received 150 mg BID of MK-8353 and 75 mg selumetinib orally with 4 days on and 3 days off until disease progression or discontinuation.
Period: Overall Study
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Started | 3 | 12 | 15
Completed | 0 | 0 | 0
Not Completed | 3 | 12 | 15
Not completed — Death | 3 | 7 | 4
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Sponsor Decision | 0 | 2 | 8
Not completed — Withdrawal by Subject | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg | Total
Number analyzed (Participants) | 3 | 12 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (8.2) | 58.6 (13.3) | 60.2 (16.1) | 59.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7 | 14
  Male | 3 | 5 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 12 | 15 | 29
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 11 | 13 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicities
Description: A dose limiting toxicity (DLT) is defined as any hematologic or non-hematologic toxicity ≥Grade 3 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. The occurrence of any of the designated toxicities during Cycle 1 (3-week cycle) were considered a DLT, if assessed by the investigator to be possibly, probably, or definitely related to study treatment administration. The number of participants experiencing DLTs was assessed.
Time Frame: Cycle 1 (3-week Cycle) (Up to 3 weeks)
Population: The analysis population included all participants who received at least 1 dose of study treatment who met the criteria for DLT evaluability (finished Cycle 1 without a DLT or experienced a DLT in Cycle 1).
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Number analyzed (Participants) | 3 | 11 | 14
Participants | 0 | 1 | 7

2. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants experiencing AEs was assessed.
Time Frame: ~90 days after last treatment dose (up to ~45 weeks)
Population: The analysis population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Number analyzed (Participants) | 3 | 12 | 15
Participants | 3 | 12 | 15

3. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants discontinuing study treatment due to AEs was assessed.
Time Frame: Up to ~33 weeks
Population: The analysis population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Number analyzed (Participants) | 3 | 12 | 15
Participants | 0 | 3 | 1

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve for MK-8353 From Time 0 to 12 Hours
Description: Blood samples were collected to determine the area under the curve from time 0 to 12 hours (AUC0-12). AUC is a measure of the amount of drug in the blood over time.
Time Frame: Study Days 1 and 4 of Cycle 1 (3-week cycle) at pre-dose and at 1, 2, 4, 6 hours, and between 8 and 12 hours post-dose
Population: The analysis population included all participants who were compliant with the study procedures and had available MK-8353 AUC data from at least 1 treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μmol/liter
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Number analyzed (Participants) | 2 | 9 | 10
hr*μmol/liter
  MK-8353, Cycle 1, Day 1 | 14.3 (62.7) | 9.66 (50.7) | 13.7 (32.8)
  MK-8353, Cycle 1, Day 4: number analyzed (Participants) | 2 | 9 | 7
  MK-8353, Cycle 1, Day 4 | 16.7 (365.7) | 19.0 (36.9) | 20.9 (60.6)

5. Secondary Outcome: AUC0-12 for Selumetinib
Description: Blood samples were collected to determine the AUC0-12. AUC is a measure of the amount of drug in the blood over time.
Time Frame: Study Days 1 and 4 of Cycle 1 (3-week cycle) at pre-dose and at 1, 2, 4, 6 hours, and between 8 and 12 hours post-dose
Population: The analysis population included all participants who were compliant with the study procedures and had available selumetinib AUC data from at least 1 treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μmol/liter
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Number analyzed (Participants) | 3 | 12 | 12
hr*μmol/liter
  Selumetinib, Cycle 1, Day 1 | 2.99 (27.2) | 5.20 (63.2) | 10.9 (49.1)
  Selumetinib, Cycle 1, Day 4: number analyzed (Participants) | 3 | 8 | 8
  Selumetinib, Cycle 1, Day 4 | 3.80 (24.6) | 6.28 (75.3) | 12.7 (31.5)

6. Secondary Outcome: Minimum Observed Plasma Concentration for MK-8353
Description: Blood samples were collected to determine the minimum observed plasma concentration (Cmin) which is the minimum amount of drug in the plasma after the dose is given. In cases where Cmin values were below the limit of quantification (BLOQ), arithmetic mean (percent coefficient of variation [%CV]) was reported instead of geometric mean (percent geometric coefficient of variation [%GCV]), since geometric mean (%GCV) was not calculable. In cases where all Cmin values were BLOQ, mean was not calculable and indicated as "NA."
Time Frame: Study Days 1 and 4 of Cycles 1 and 2 (3-week cycles). For Cycle 1, pre-dose and at 1, 2, 4, 6 hours, and between 8 and 12 hours post-dose; and for Cycle 2 pre-dose, and at 1 and 4 hours post-dose
Population: The analysis population included all participants who were compliant with the study procedures and had available MK-8353 Cmin data from at least 1 treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/liter
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Number analyzed (Participants) | 3 | 10 | 13
μmol/liter
  MK-8353, Cycle 1, Day 1: number analyzed (Participants) | 3 | 10 | 11
  MK-8353, Cycle 1, Day 1 | NA (NA) — NA=All Cmin values of MK-8353 plasma concentrations were BLOQ at Cycle 1 Day 1 and Geometric Mean (%GCV) was not calculable. | NA (NA) — NA=All Cmin values of MK-8353 plasma concentrations were BLOQ at Cycle 1 Day 1 and Geometric Mean (%GCV) was not calculable. | NA (NA) — NA=All Cmin values of MK-8353 plasma concentrations were BLOQ at Cycle 1 Day 1 and Geometric Mean (%GCV) was not calculable.
  MK-8353, Cycle 1 Day 4: number analyzed (Participants) | 3 | 8 | 13
  MK-8353, Cycle 1 Day 4 | 0.695 (222.6) | 1.10 (50.6) | 1.47 (455.5)
  MK-8353, Cycle 2 Day 1: number analyzed (Participants) | 3 | 10 | 11
  MK-8353, Cycle 2 Day 1 | 0.0361 (173.2) | 0.0313 (191.0) | 0.0166 (189.7)
  MK-8353, Cycle 2 Day 4: number analyzed (Participants) | 3 | 9 | 11
  MK-8353, Cycle 2 Day 4 | 0.598 (172.6) | 0.995 (90.7) | 1.47 (84.8)

7. Secondary Outcome: Cmin for Selumetinib
Description: Blood samples were collected to determine the Cmin which is the minimum amount of drug in the plasma after the dose is given. In cases where Cmin values were BLOQ, arithmetic mean (%CV) was reported instead of geometric mean (%GCV), since geometric mean (%GCV) was not calculable. In cases where all Cmin values were BLOQ, mean was not calculable and indicated as "NA."
Time Frame: as for outcome 6
Population: The analysis population included all participants who were compliant with the study procedures and had available selumetinib Cmin data from at least 1 treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/liter
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Number analyzed (Participants) | 3 | 10 | 11
μmol/liter
  Selumetinib, Cycle 1, Day 1: number analyzed (Participants) | 3 | 10 | 10
  Selumetinib, Cycle 1, Day 1 | NA (NA) — NA=All Cmin values of Selumetinib plasma concentrations were BLOQ at Cycle 1 Day 1 and Geometric Mean (%GCV) was not calculable. | NA (NA) — NA=All Cmin values of Selumetinib plasma concentrations were BLOQ at Cycle 1 Day 1 and Geometric Mean (%GCV) was not calculable. | NA (NA) — NA=All Cmin values of Selumetinib plasma concentrations were BLOQ at Cycle 1 Day 1 and Geometric Mean (%GCV) was not calculable.
  Selumetinib, Cycle 1, Day 4: number analyzed (Participants) | 3 | 8 | 11
  Selumetinib, Cycle 1, Day 4 | 0.101 (35.1) | 0.265 (38.9) | 0.456 (160.1)
  Selumetinib, Cycle 2, Day 1: number analyzed (Participants) | 3 | 10 | 10
  Selumetinib, Cycle 2, Day 1 | NA (NA) — NA=All Cmin values of Selumetinib plasma concentrations were BLOQ at Cycle 2 Day 1 and Geometric Mean (%GCV) was not calculable. | 0.00202 (232.9) | 0.00124 (215.7)
  Selumetinib, Cycle 2, Day 4: number analyzed (Participants) | 3 | 9 | 10
  Selumetinib, Cycle 2, Day 4 | 0.127 (74.6) | 0.174 (80.3) | 0.257 (47.5)

8. Secondary Outcome: Maximum Observed Plasma Concentration for MK-8353
Description: Blood samples were collected to determine the maximum observed plasma concentration (Cmax) which is the measure of the maximum amount of drug in the plasma after the dose is given.
Time Frame: Study Days 1 and 4 of Cycle 1 (3-week cycle) at pre-dose and at 1, 2, 4, 6 hours, and between 8 and 12 hours post-dose
Population: The analysis population included all participants who were compliant with the study procedures and had available MK-8353 Cmax data from at least 1 treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/liter
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Number analyzed (Participants) | 3 | 12 | 15
μmol/liter
  MK-8353, Cycle 1, Day 1 | 1.24 (138.4) | 1.65 (60.9) | 2.95 (62.3)
  MK-8353, Cycle 1, Day 4: number analyzed (Participants) | 3 | 10 | 13
  MK-8353, Cycle 1, Day 4 | 1.87 (149.4) | 2.53 (51.5) | 3.61 (80.9)

9. Secondary Outcome: Cmax for Selumetinib
Description: Blood samples were collected to determine the Cmax which is the measure of the maximum amount of drug in the plasma after the dose is given.
Time Frame: Study Days 1 and 4 of Cycle 1 (3-week cycle) at pre-dose and at 1, 2, 4, 6 hours, and between 8 and 12 hours post-dose
Population: The analysis population included all participants who were compliant with the study procedures and had available selumetinib Cmax data from at least 1 treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/liter
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
Number analyzed (Participants) | 3 | 12 | 13
μmol/liter
  Selumetinib, Cycle 1,Day 1 | 1.01 (29.7) | 1.96 (91.1) | 3.37 (57.1)
  Selumetinib, Cycle 1, Day 4: number analyzed (Participants) | 3 | 10 | 11
  Selumetinib, Cycle 1, Day 4 | 1.04 (13.3) | 1.44 (123.6) | 2.37 (107.5)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (NSAEs): Up to ~45 weeks; Serious adverse events (SAEs): Up to ~45 weeks. All-cause mortality: Up to 24 months
Description: NSAE, SAE, and all-cause mortality tables include all randomized participants who received at least 1 dose of study drug. Per protocol, disease progression of cancer was not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | MK-8353 50 mg + Selumetinib 25 mg | MK-8353 100 mg + Selumetinib 50 mg | MK-8353 150 mg + Selumetinib 75 mg
All-Cause Mortality (participants affected / at risk) | 3/3 | 8/12 | 6/15
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/12 | 4/15
Other Adverse Events (participants affected / at risk) | 3/3 | 11/12 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8353 50 mg + Selumetinib 25 mg (N=3) | MK-8353 100 mg + Selumetinib 50 mg (N=12) | MK-8353 150 mg + Selumetinib 75 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8353 50 mg + Selumetinib 25 mg (N=3) | MK-8353 100 mg + Selumetinib 50 mg (N=12) | MK-8353 150 mg + Selumetinib 75 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 2 (4)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 7 (9) | 12 (25)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (7) | 7 (10)
Oral pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4) | 4 (8)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 8 (11)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 4 (5)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT03745989/Prot_SAP_000.pdf